CLINICAL TRIAL: NCT02879760
Title: A Phase 1/2 Trial of MG1 Maraba Expressing MAGE-A3 (MG1-MAGEA3), With Adenovirus Vaccine Expressing MAGE-A3 (Ad-MAGEA3), in Combination With Pembrolizumab in Patients With Previously Treated Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Oncolytic MG1-MAGEA3 With Ad-MAGEA3 Vaccine in Combination With Pembrolizumab for Non-Small Cell Lung Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Turnstone Biologics, Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ad/MG1-MAGEA3-001 (Sandpiper)
Record Dates: First submitted 2016-08-15; First posted 2016-08-26 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Lung; Cancer; Chemotherapy; Oncolytic virus; Immunotherapy; Pembrolizumab; Keytruda
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ad/MAGEA3, MG1-MAGEA3 and pembrolizumab (Experimental): Ad-MAGEA3 prime will be administered as a single IM dose on Day 1 at 2 x 10e11 VP.
  MG1/MAGEA3 boost will be administered IV on Day 15 and Day 18 by 5 cohorts: Cohort 1: Days 15 & 18 at 1x 10e10 pfu.
  Cohort 2: Days 15 & 18 at 1x 10e11 pfu. Cohort 3: Day 15 at 1 x 10e11 pfu; Day 18 at 3 x 10e11 pfu. Cohort 4: Day 15 at 1 x 10e11 pfu; Day 18 at 3 x 10e11 pfu. Cohort 5: Day 15 at 3x 10e11 pfu; Day 18 at 3 x 10e12 pfu. Pembrolizumab will be administered IV every 3 weeks starting on Day 22.
  Interventions: Biological: Ad-MAGEA3; Biological: MG1-MAGEA3; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Ad-MAGEA3 — Intramuscular injection
Biological: MG1-MAGEA3 — Intravenous infusion
Biological: Pembrolizumab — Intravenous infusion

SUMMARY:
This is a Phase 1/2, multi-center, open-label, dose-escalation trial of Ad-MAGEA3 and MG1-MAGEA3 in combination with pembrolizumab in patients with Non-Small Cell Lung Cancer who have completed a first standard therapy with at least 1 cycle of platinum based chemotherapy and/or at least one treatment of PD-1 or PD-L1 antibody targeted therapy.

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, dose-escalation trial of Ad MAGEA3 and MG1-MAGEA3 in combination with pembrolizumab in patients with NSCLC (histological subtype of squamous and non-squamous NSCLC). In Phase 1, patients who have progressed after treatment with a platinum-based regimen and/or PD-1/PD-L1 targeted antibody therapy will be enrolled. In Phase 2, only patients who have progressed after treatment regimen containing PD-1/PD-L1 targeted antibody therapy will be enrolled. In the Phase 1 portion of the study, MG1-MAGEA3 treatment will be escalated in a sequential dose-escalating design. In the Phase 2 portion of the study, MG1-MAGEA3 treatment will be at the maximum tolerated dose (MTD) or the maximum feasible dose (MFD). The Ad-MAGEA3 and pembrolizumab dose is fixed in both the Phase 1 and Phase 2 portions of the trial.

Phase 1 Enrollment

Cohorts 1 through 5:

Three patients will be treated at each dose level unless a dose-limiting toxicity (DLT), as defined below, is observed. Patients will be observed for a DLT through Day 29. After enrollment of the first patient in each cohort, 2 additional patients will be enrolled after the initial patient reaches Day 29 without experiencing a DLT. Treatment with MG1-MAGEA3 will proceed to the next dose level if 0 of 3 patients experiences a DLT. If one of the first 3 patients experiences a DLT, additional patients will be enrolled until a second patient experiences a DLT (which defines the toxic dose) or until 6 total patients have been treated, whichever comes first. If a second DLT is not experienced within that cohort, dose escalation may continue.

If 2 DLTs are observed within a cohort, enrollment into the cohort will cease and the dose level immediately preceding that dose will be determined as the MTD.

Ad-MAGEA3 will be administered by intramuscular (IM) injection at a dose level of 2 x 1011 virus particles (VP) on Day 1. MG1-MAGEA3 will be administered by intravenous (IV) infusion at escalating dose levels on Day 15 and Day 18. In Cohorts 1 through 5, patients will receive pembrolizumab at a dose of 200 mg IV on Day 22, and every 3 weeks thereafter until confirmed radiographic progression or unmanageable toxicity.

Cohort 6:

Upon determination of the MTD/MFD (safety assessment) in Cohorts 4-5, the treatment regimen will next be optimized such that pembrolizumab will begin on Day 1 (concurrent treatment). The Day 15 and Day 18 doses of MG1-MAGEA3 will be the doses defined as the MTD/MFD in either Cohort 4 or5. Specifically, the regimen evaluated in Cohort 6 is as follows:

* Day 1: Patients will receive 2 x 1011 VP IM of Ad-MAGEA3 and 200 mg IV of pembrolizumab (the Pembrolizumab will be continued every 3 weeks [Q3W]).
* Day 15: Patients will receive IV MG1-MAGEA3 at the MTD/MFD established for the first infusion from Cohort 4 or Cohort 5.
* Day 18: Patients will receive IV MG1-MAGEA3 at the MTD/MFD established for the second infusion from Cohort 4 or Cohort 5.
* Three patients will be treated according to the dose schedule above unless a DLT is observed between Day 1 and Day 29, at which time three additional patients will be enrolled onto this cohort. If 2 DLTs occur within these six patients treated in Cohort 6, this cohort will be stopped and a new Cohort will be initated again with patients treated concurrently with pembrolizumab but with a 0.5 log lower dose of MG1-MAGEA3 than used in Cohort 6 for the Day 15 and Day 18 doses.

Phase 2 Enrollment Phase 2 enrollment will commence upon completion of dose escalation and determination of the MTD/MFD. In Stage 1 of the 2-Stage design, 18 evaluable patients will be treated at the MTD/MFD (this will include patients treated at the MTD/MFD in Phase 1 who meet Phase 2 inclusion criteria). If 1 or more patients respond, the study may continue to Stage 2, and an additional 14 evaluable patients will be enrolled for a total of 32 evaluable patients.

A patient will be defined as being evaluable for the primary endpoint (EPPE) and included in the Simon 2-stage study design if they are seronegative to adenovirus Type 5, the virus used in the prime.

Preliminary data from two other Turnstone Ad/MG1-MAGEA3 trials indicates that patients without pre-existing anti-adenovirus antibodies (seronegative) prior to treatment have a greater likelihood of generating MAGEA3 specific T-cell responses than those that are seropositive at baseline. Therefore, this study is designed to primarily determine the response rate and clinical outcome for this homogenous population of Ad5 seronegative patients whom are most likely to benefit from Ad/MG1-MAGEA3 treatment. However, there is a small subset of seropositive patients who developed significant anti-MAGEA3 T-cell responses after Ad/MG1-MAGEA3 treatment. In addition, the presence of Ad5 seropositivity would not be expected to have any significant impact on the potential benefit of MG1-MAGEA3 tumor oncolysis. Therefore, exploratory data on clinical and immune response in the Ad5 seropositive population will be conducted and the study will enroll both Ad5 seronegative and positive patients.

It is anticipated that approximately half of the patients enrolled will be seronegative to Ad5, therefore Stage 1 of the Simon 2-stage design above will enroll approximately 18 patients and Stage 2 will enroll approximately 14 patients. Total study enrollment is projected to be between 2 and 100 patients.

Safety Committee:

Prior to each dose level increase or the initiation of Phase 2, a safety committee composed of independent voting members and treating physician(s) will review toxicity and other relevant data to determine suitability of dose escalation or expansion with regards to patient safety. Interim assessments of toxicity will be conducted throughout the trial to monitor for safety trends and identify any new or increased toxicity not previously associated with the IPs.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the patient must:

1. Have histologically or cytologically confirmed diagnosis of NSCLC (squamous or non-squamous) with positive expression of MAGE-A3 (primary or metastatic lesion).
2. Phase 1: Have radiographic progression after treatment with at least 1 cycle of platinum-doublet chemotherapy and/or at least one treatment of PD-1 or PD-L1 antibody targeted therapy. Adjuvant therapy will count as a regimen if administered within 1 year before relapse.

   Phase 2: Have radiographic progression during or after treatment with anti-PD-1/PD-L1 antibody. Adjuvant therapy will count as regimen if administered within 1 year before relapse.
3. Phase 1: Patients with tumors of non-squamous NSCLC histology that have a known epidermal growth factor receptor (EGFR) mutation and/or anaplastic lymphoma kinase (ALK) translocation can participate in the Phase 1 portion of the study if they have failed the appropriate tyrosine kinase inhibitor (TKI) (intolerance or documented progression of their NSCLC) and have documented progression of their NSCLC. There is no preferred order of treatment with TKI or platinum doublet therapy. If a patient is found to have one molecular alteration (either sensitizing EGFR mutation or ALK translocation), then testing for the other alteration is not required.

   Phase 2: Patients with the above ALK and EGFR targetable mutations will not be eligible for treatment.
4. Have measurable disease based on RECIST v1.1 criteria as determined by the site study team. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions post irradiation treatment.
5. Have at least one tumor amenable to biopsy.
6. Have Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Demonstrate adequate organ function:

   1. White blood cell (WBC) count ≥3,000 cells/mm3
   2. Absolute neutrophil count (ANC) ≥1,000 cells/mm3
   3. Hemoglobin ≥8 g/dL or ≥4.96 mmol/L (correction with transfusion or erythropoietin-based therapy allowed to meet eligibility criteria)
   4. Platelet count ≥100,000 platelets/mm3 (untransfused)
   5. Total bilirubin ≤1.5 x Upper Limit of Normal (ULN) OR direct bilirubin ≤ULN for patients with total bilirubin levels >1.5 x ULN (i.e., patients with Gilberts disease)
   6. Aspartate transaminase (AST), alanine aminotransferase (ALT) ≤2.5 x ULN; ≤5.0 x ULN if patient has liver metastases
   7. Serum chemistries Sodium, Potassium, and Calcium within normal limits (WNL) or Grade 1
   8. Serum creatinine ≤1.5 x ULN or creatinine clearance ≥60 mL/min for patient with creatinine levels >1.5 institutional ULN according to Cockcroft-Gault formula
   9. Serum phosphate >0.8 mmol/L (Grade 0-1)
   10. International normalized ratio (INR) ≤1.5 x ULN unless patient is receiving anticoagulant therapy as long as prothrombin time (PT) or partial prothrombin time (PTT) is within therapeutic range of intended use of anticoagulants
   11. Activated partial thromboplastin time (aPTT) ≤1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
   12. Resting oxygen saturation on room air ≥ 90%
8. Female patients of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female patients of childbearing potential (refer to Section 11.A.2.c) must be willing to use an adequate method of contraception as outlined in Section 11.A.2.c, starting with Day 1 through 120 days after the last dose of study medication.

   Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.
10. Male patients of reproductive potential (Section 11.A.2.c) must agree to use an adequate method of contraception as outlined in Section 11.A.2.c, starting with Day 1 through 120 days after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.
11. Be willing and able to provide written informed consent for the trial.
12. Be 18 years of age (or legal age of majority in the jurisdiction) on day of signing informed consent.

Exclusion Criteria:

The patient must be excluded from participating in the trial if the patient:

1. Has disease that is suitable for local therapy administered with curative intent.
2. Has had prior treatment with any MAGE-A3 vaccine immunotherapy including Ad-MAGEA3 or MG1-MAGEA3.
3. Is currently receiving experimental therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
4. Has had prior anti-cancer monoclonal antibody (mAb) therapy within 4 weeks prior to study Day 1 or failure to recover (i.e., to ≤ Grade 1 or to baseline status) from adverse events (AEs) due to agents administered more than 4 weeks earlier.
5. Has been intolerant of prior PD-1/PD-L1 targeted antibody therapy for which re-treatment would expose the patient to clinically significant risk in the opinion of the investigator (please attain sponsor permission of enrollment of any patient with prior intolerance to anti-PD-1/PD-L1 antibody treatment).
6. Has had prior chemotherapy, or targeted small molecule therapy, or radiation therapy within 4 weeks prior to study Day 1 or who has not recovered (i.e., to ≤ Grade 1 or to baseline status) from AEs due to a previously administered agent.

   Note: Patients with ≤Grade 2 neuropathy or having any alopecia are an exception to this criterion and may qualify for the study.

   Note: If patient received major surgery, they must be at least 4 weeks from surgery AND have recovered adequately from the toxicity and/or complications from the surgery prior to starting therapy.

   Note: Patients receiving prior radiation must have recovered (< Grade 1) from any acute toxicity. Patients having irreversible but not clinically significant toxicity are eligible.

   Note: Patients receiving prior lung radiation with a dose of >30 Gy must wait at least 8 weeks from the date of completion of the lung radiation before the first dose of pembrolizumab.
7. Has received prior treatment with vesicular stomatitis virus (VSV) based viral vector.
8. Requires use of anti-platelet or anti-coagulant therapy that cannot be safely suspended for per protocol biopsies as per standard of care.
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.

   Note: Patients with previously treated brain metastases who are stable may participate. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
10. Has clinically significant tumor invasion (e.g., impeding obstruction) of a major vascular structure (e.g., carotid artery) or other key anatomical structure (e.g., pulmonary airway) or clinically significant and/or rapidly accumulating ascites, pericardial or pleural effusions.
11. Has active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Has evidence of active, non-infectious pneumonitis or current radiographic evidence of pneumonitis.
13. Has a history of interstitial lung disease.
14. Has an active infection requiring systemic therapy.
15. Has known active Hepatitis B (e.g., Hepatitis B surface antigen [HBsAg] reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected) virus infection.
16. Has used anti-viral medication, within 14 days of enrollment.
17. Has conditions likely to have resulted in splenic dysfunction (e.g., splenectomy, sickle cell anemia, radiation to the spleen >20 Gy, congenital asplenism).
18. Has significant immunodeficiency due to underlying illness (e.g., known HIV/AIDS).
19. Has received immunosuppressive medication (e.g., systemic corticosteroids) within 4 weeks prior to the first dose of trial treatment.

    Note: Patients must not be receiving doses of >10 mg/day of prednisone or equivalent at the time of study entry and corticosteroids may not be used for premedication.
20. Previous solid organ or allogeneic stem cell transplant.
21. Has uncontrolled pre-existing cardiovascular conditions and/or symptomatic cardiac dysfunction.
22. Has >Grade 2 dyspnea and/or requirement for supplemental oxygen.
23. Has received a live vaccine within 30 days of planned start of study therapy (Note: killed flu vaccine acceptable).
24. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
25. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
26. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
27. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with Day 1 through 120 days after the last dose of study medication (including pembrolizumab).
28. History of severe allergic anaphylactic reactions to chimeric, human or humanized antibodies, or fusion proteins.
29. Patients with household contacts meeting any of the following criteria for study entry unless alternate living arrangements can be made, while under contact precautions (from the time of initial treatment with MG1-MAGEA3 until at least 7 days after the last dose of MG1-MAGEA3):

    1. Women who are pregnant or nursing an infant
    2. Children <1 year old; or
    3. Individuals who are severely immunocompromised (including but not limited to: bone-marrow or organ transplant recipients; individuals with human Immunodeficiency virus [HIV] infection; individuals receiving chronic immunosuppressive medication such as systemic corticosteroids).
30. Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or Sponsor staff directly involved with this trial, unless prospective IRB approval (by chair or designee) is given allowing exception to this criterion for a specific patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-05-24 (Actual)

PRIMARY OUTCOMES:
Phase 1 - Toxicity as measured by adverse events | 7 months
  To determine the maximum tolerated dose MTD/ maximum feasible dose MFD of Ad/MAGEA3 and MG1-MAGEA3 in combination with pembrolizumab
Phase 2 - Objective tumour response rate (ORR) based on RECIST v1.1 | 7 months
  To evaluate objective tumour response rate (ORR) based on RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Breitbach, PhD, Study Director — Turnstone Biologics, Corp.
Locations (6):
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Moncton Hospital, Moncton, New Brunswick
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jenner AL, Cassidy T, Belaid K, Bourgeois-Daigneault MC, Craig M. In silico trials predict that combination strategies for enhancing vesicular stomatitis oncolytic virus are determined by tumor aggressivity. J Immunother Cancer. 2021 Feb;9(2):e001387. doi: 10.1136/jitc-2020-001387. PMID 33608375
- [Derived] Pol JG, Acuna SA, Yadollahi B, Tang N, Stephenson KB, Atherton MJ, Hanwell D, El-Warrak A, Goldstein A, Moloo B, Turner PV, Lopez R, LaFrance S, Evelegh C, Denisova G, Parsons R, Millar J, Stoll G, Martin CG, Pomoransky J, Breitbach CJ, Bramson JL, Bell JC, Wan Y, Stojdl DF, Lichty BD, McCart JA. Preclinical evaluation of a MAGE-A3 vaccination utilizing the oncolytic Maraba virus currently in first-in-human trials. Oncoimmunology. 2018 Sep 19;8(1):e1512329. doi: 10.1080/2162402X.2018.1512329. eCollection 2019. PMID 30546947